CLINICAL TRIAL: NCT03410797
Title: Efficacy of a Semi-occluded Mask in the Treatment of Patients With Voice Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacqueline Gartner-Schmidt (Other)
Responsible Party: Sponsor-Investigator, Jacqueline Gartner-Schmidt, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO17100675
Record Dates: First submitted 2018-01-05; First posted 2018-01-25 (Actual); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Voice and Resonance Disorders; Vocal Fold Polyp; Vocal Cord Cyst; Vocal Cord Polyp; Atrophy of Vocal Cord
Keywords: SOVT; semi occluded vocal tract; voice disorder; voice therapy; muscle tension dysphonia; MTD; vocal fold lesions; vocal fold atrophy
MeSH Terms: conditions — Voice Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Voice Disorder Requiring Voice Therapy (Other): Individuals with a voice disorder such as muscle tension dysphonia (MTD), vocal fold atrophy or vocal fold lesions recommended for voice therapy as treatment.
  Interventions: Device: Inclusion of semi-occluded mask in voice therapy

INTERVENTIONS:
Device: Inclusion of semi-occluded mask in voice therapy — Patients will be given a facemask with a semi-occlusion (SOMask) for use during in person voice therapy and for use at home therapy practice.

SUMMARY:
Current semi-occluded vocal tract therapies limit the type of vocalizations that can be produced to single vowels, which does not promote learning of the healthy voice behavior in connected speech or generalization to conversation. However, recent preliminary results using a semi-occluded mask indicate that the use of certain mask port diameters may allow for natural speech production while increasing supraglottal pressure and impedance, and thereby result in elicitation of voice with increased efficiency. In addition, the use of a semi-occluded mask provides the possibility for a better transition from phonating single phonemes in therapy to training the target therapy techniques in connected speech.

DETAILED DESCRIPTION:
Treatment of voice disorders varies but often involves voice therapy and/or surgical intervention. Voice therapy, a non-invasive behavioral treatment for voice disorders, helps patients develop beneficial voice habits, prevents recurrence of voice disorders, and facilitates long-lasting vocal improvement. Many voice therapy techniques involve a semi-occluded vocal tract (SOVT). SOVT treatment is often characterized by sustained (straw phonation, voiced fricatives, nasals), oral oscillatory (lip buzzes, tongue trills, raspberries) or transitory phonation (plosives and glides). Straw phonation therapy, one of the most utilized SOVT methods, was first proposed in 1904 and involved phonating at different pitches into small glass tubes with varying diameters and lengths providing simultaneous semi-occlusion and extension of the vocal tract. Voice therapy exercises involving voice production with a semi-occluded and sometimes lengthened vocal tract have demonstrated improved vocal efficiency and loudness, reduced mechanical trauma to the vocal fold mucosa, and improved source-filter interaction.Our group recently developed a semi-occluded facemask for use in patients with and without voice disorders. Recent preliminary results using this semi-occluded facemask indicated that the use of a certain mask port diameters may elicit voice with increased efficiency. A study of 5 participants without voice disorders revealed that a mask occlusion diameter of 6.4 and 3.2 mm resulted in improved vocal efficiency. A study of the immediate effects of a semi-occluded facemask in 20 patients with voice disorders revealed that occlusions diameters of 9.6, 6.4, and 3.2 mm all resulted in significant improvements in acoustic and aerodynamic voice outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 60
* diagnosed with vocal fold lesion or polyp or cyst or atrophy or other voice condition (such as muscle tension dysphonia)
* recommended for voice therapy as treatment for voice disorder

Exclusion Criteria:

* Current smoker (greater than 5 cigarettes/week)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Any data shared would be completely de-identified. Currently there is no plan to share information at this time.
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: additional researchers may receive de-identified information only if a data use agreement has been executed.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Voice Disorder Requiring Voice Therapy
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Voice Disorder Requiring Voice Therapy
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 38 [19 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 11
Voice Handicap Index - 10 [Mean (Full Range); unit: units on a scale] — This is a self report questionnaire describing the quality of voice problems. Consists of 10 questions. Each question has a minimum value of 0 and a maximum value of 4.
  A score of 0 is the lowest overall score. A score of 40 is the maximum overall score.
  The higher the value, the greater the voice problem.
  units on a scale | 17 [12 to 34]
Cepstral Peak Prominance-CPP [Mean (Full Range); unit: decibels] — an objective, acoustic measure of voice quality that has been qualified as a robust acoustic measure of dysphonia severity
  decibels | 10.43 [5.7 to 14.83]
Cepstral Spectral Index of Dysphonia (CSID) [Mean (Full Range); unit: units on a scale] — CSID is an objective evaluation of voice recordings through specialized vocal analysis software.
  The CSID is a multifactorial estimate of vocal severity that correlates with the labeled visual analog scale for severity (in %). Normal cutoff range is from 19-24. Values outside of this range are considered to have varying degrees of dysphonia. The values are captured using specialized voice analysis equipment and analyzed using the specialized CSID software. CSID can be calculated as both negative and positive integers with no true boundaries
  units on a scale | -3.46 [-13.51 to 66.15]
Mean Airflow [Mean (Full Range); unit: mL/s] — Aerodynamic measure of airflow. Increased airflow leads to better voice mechanics and better voice quality.
  mL/s | 138 [66 to 291]
Mean vocal intensity [Mean (Full Range); unit: dB SPL] — Acoustic measure of voice
  dB SPL | 66.75 [61.28 to 73.52]
Voice Diagnoses [Number; unit: participants]
  Diagnosis of Lesions | 3
  Diagnosis of Muscle Tension Dysphonia | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in VHI-10 Score After 4 Sessions of Voice Therapy
Description: VHI-10 is a 10 item, self reported, voice related outcome related to an individual's perception of their vocal quality and how it impacts their life. (Voice Handicap Index) Scale scores range from 0-40 where higher scores correspond to a worse vocal quality.
Time Frame: Baseline and approximately 6-8 weeks later; after completion of voice therapy
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | Voice Disorder Requiring Voice Therapy
Number analyzed (Participants) | 11
score on a scale | 7 [-3 to 17]
Statistical Analysis 1: Comparison: Voice Disorder Requiring Voice Therapy; Descriptive statistics characterized this patient perception measurement; Test type: Other — Due to small sample size, nonparametric Wilcoxon signed-rank tests were used to compare VHI-10 before and after therapy; p = .0076, Wilcoxon (Mann-Whitney); Median Difference (Net) = 7

2. Secondary Outcome: Change From Baseline in Cepstral Peak Prominence (dB)
Description: CPP is an objective evaluation of voice recordings through specialized vocal analysis software.
Time Frame: Baseline and approximately 6-8 weeks later; after completion of voice therapy
Measure: Median (95% Confidence Interval); unit: dB
Groups:
- Voice Disorder Requiring Voice Therapy: Individuals with a voice disorder such as muscle tension dysphonia (MTD), vocal fold atrophy or vocal fold lesions recommended for voice therapy as treatment.
  Inclusion of semi-occluded mask in voice therapy: Patients will be given a facemask with a semi-occlusion (SOMask) for use during in person voice therapy and for use at home therapy practice.
  Three of the subjects carried a diagnosis of lesions and 8 subjects carried a diagnosis of muscle tension dysphonia.
Arm/Group | Voice Disorder Requiring Voice Therapy
Number analyzed (Participants) | 11
dB | -1.53 [-9.60 to 1.17]
Statistical Analysis 1: Comparison: Voice Disorder Requiring Voice Therapy; Test type: Other — Descriptive statistics characterized acoustic and aerodynamic measures, and patient perception measurements; p = .0329, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -1.53

3. Secondary Outcome: Change From Baseline in Cepstral Spectral Index of Dysphonia (CSID--a Multivariate Estimate of Dysphonia Severity)
Description: CSID is an objective evaluation of voice recordings through specialized vocal analysis software.
  The CSID is a multifactorial estimate of vocal severity that correlates with the labeled visual analog scale for severity (in %). Normal cutoff range is from 19-24. Values outside of this range are considered to have varying degrees of dysphonia. The values are captured using specialized voice analysis equipment and analyzed using the specialized CSID software.
  Depending on the voice disorder, CSID can be calculated as both negative and positive integers with no true boundaries.
Time Frame: Baseline and approximately 6-8 weeks later; after completion of voice therapy
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Voice Disorder Requiring Voice Therapy
Number analyzed (Participants) | 11
units on a scale | 15.39 [-6.92 to 81.95]
Statistical Analysis 1: Comparison: Voice Disorder Requiring Voice Therapy; Test type: Other — Descriptive statistics characterized acoustic and aerodynamic measures, and patient perception measurements; p = .0164, Wilcoxon (Mann-Whitney); Median Difference (Net) = 15.39

4. Secondary Outcome: Change From Baseline in Mean Airflow in Milliliters (ml) During Reading of Standardized Paragraph
Description: mean airflow will be captured during the phonatory aerodynamic system (PAS) recording of airflow during the reading of the standardized paragraph.
Time Frame: Baseline and approximately 6-8 weeks later; after completion of voice therapy
Measure: Median (95% Confidence Interval); unit: milliliters
Arm/Group | Voice Disorder Requiring Voice Therapy
Number analyzed (Participants) | 11
milliliters | -52 [-138 to 105]
Statistical Analysis 1: Comparison: Voice Disorder Requiring Voice Therapy; Test type: Other — Descriptive statistics characterized acoustic and aerodynamic measures, and patient perception measurements; p = 0.1141, Wilcoxon (Mann-Whitney); Median Difference (Net) = -52

5. Secondary Outcome: Change From Baseline in Mean Vocal Intensity (dB)
Description: mean vocal intensity will be captured during the phonatory aerodynamic system (PAS) recording of airflow during the reading of the standardized paragraph.
Time Frame: Baseline and approximately 6-8 weeks later; after completion of voice therapy
Measure: Median (95% Confidence Interval); unit: decibels
Arm/Group | Voice Disorder Requiring Voice Therapy
Number analyzed (Participants) | 11
decibels | -1.7 [-19.11 to 6.44]
Statistical Analysis 1: Comparison: Voice Disorder Requiring Voice Therapy; Test type: Other — Descriptive statistics characterized acoustic and aerodynamic measures, and patient perception measurements; p = .3329, Wilcoxon (Mann-Whitney); Median Difference (Net) = -1.70

6. Secondary Outcome: Change in the Number of Breaths Taken During Reading of Standardized Paragraph
Description: Numeric value of the number of breaths needed to complete the reading of a paragraph.
  Values are positive integers
Time Frame: Baseline to post treatment
Population: This information was not collected during this study on any of the participants. Therefore, there was no data to analyze.
Arm/Group | Voice Disorder Requiring Voice Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: approximately 6 weeks for each participant
Arm/Group | Voice Disorder Requiring Voice Therapy
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: Study Protocol with Statistical Analysis Plan (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/97/NCT03410797/Prot_SAP_001.pdf